CLINICAL TRIAL: NCT01655290
Title: Single Dose Gadobutrol in Comparison to Single Dose Gadobenate Dimeglumine for Magnetic Resonance Imaging of Chronic Myocardial Infarction at 3 Tesla
Brief Title: Comparison of Gadobutrol and Gadobenate Dimeglumin for Delayed Enhancement Cardiac MRI
Acronym: Gadovit
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: GAD-1140-WIL-0020-I
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Subacute/Chronic Myocardial Infarction
MeSH Terms: interventions — gadobutrol; gadobenic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gadobutrol (Experimental): first session gadobutrol second session gadobenate dimeglumin
  Interventions: Other: Gadovist® (Gadobutrol), Multihance® (Gadobenate dimeglumin)
- Demeglumin (Experimental): first session gadobenate dimeglumin second session gadobutrol
  Interventions: Other: Gadovist® (Gadobutrol), Multihance® (Gadobenate dimeglumin)

INTERVENTIONS:
Other: Gadovist® (Gadobutrol), Multihance® (Gadobenate dimeglumin) — Other (Diagnostic)

SUMMARY:
This study aims at evaluating the diagnostic efficacy of Gadobutrol versus Gadobenate dimeglumine at similar dose of 0.1mmol/kg for assessment of myocardial infarction by delayed enhancement cardiac Magnetic Resonance Imaging

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myocardial infarction
* Age ≥ 18 years and ≤ 80 years
* Informed consent
* Male patients as well as female patients using contraceptives

Exclusion Criteria:

* Patients with a heart pacemaker, with magnetic material or other magnetic implants.
* Renal failure (GFR <30ml/min)
* Patients with known allergy to a Gadolinium-containing contrast agent
* Drugs or alcohol addiction, dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Efficacy (contrast-to-noise ratio)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Radiologie - Klinikum Rechts der Isar, Munich, Bavaria, Germany